CLINICAL TRIAL: NCT00403104
Title: A Multi-centre, Randomized, Double Blind, Placebo-controlled, Parallel Group Study to Investigate Efficacy and Safety of ONO-2506PO Compared to Placebo, in the Presence of Riluzole, to Patients Diagnosed With Amyotrophic Lateral Sclerosis (ALS), Who Have Had Onset of Muscle Weakness Within 14 Months of Randomization
Brief Title: Placebo Controlled Study of ONO2506PO in the Presence of Riluzole in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-2506POE014
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: ONO-2506PO; Amyotrophic Lateral Sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- E (Experimental): ONO-2506PO in the presence of Riluzole
  Interventions: Drug: ONO-2506PO
- P (Placebo Comparator): Placebo in the presence of Riluzole
  Interventions: Drug: ONO-2506PO

INTERVENTIONS:
Drug: ONO-2506PO — 1200 mg QD / 18 months
  Arms: E
Drug: ONO-2506PO — 0 mg QD / 18 months
  Arms: P

SUMMARY:
The purpose of this study is to determine if oral treatment with ONO-2506PO in patients diagnosed with ALS, who have had onset of muscle weakness within 14 months of randomization, could lead to the slowing of decline in respiratory function, functional status, muscle strength, quality of life and survival compared with placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of clinically possible, clinically probable laboratory-supported, clinically probable or clinically definite ALS (according to WNF EL Escorial diagnostic criteria, revised according to the Airlie House Conference 1998)
2. Onset of muscle weakness within 14 months randomization
3. Concomitant standard Riluzole therapy (50mg twice daily)

Exclusion Criteria:

1. Presence of a tracheotomy, mechanical ventilation or non-invasive ventilation
2. Requirement for prescription drugs used for potential neuroprotective benefit -

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Rate of decline of respiratory function determined as SVC over the 12 month treatment period | 12 months

SECONDARY OUTCOMES:
Survival | 12, 18 months
Functional Assessment (ALSFRS-R) | 12, 18 months
Muscle Strength (MRC muscle score) | 12, 18 months
Quality of Life | 12, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Tomohiro Kuwayama, Study Director — Ono Pharmaceutical Co. Ltd
Locations (26):
- L. Boltzmann Forschungsinstitut, Neurologische Abteilung, Kaiser Franz Josef Hospital, Wien, Vienna, Austria
- Belgium (2):
  - UCL Saint-Luc, Brussels
  - UZ Leuven, Leuven
- France (6):
  - Hopital Roger Salengro - Clinique Neurologique, Neurologie A, Lille
  - Hopital Duruytren, Limoges
  - Hopital de la Timone, Marseille
  - Hopital de Chauliac, Montpellier
  - Hopital l-Archet 1, Nice
  - Hopital LaPitie Salpetriere, Paris
- Germany (8):
  - Charite Campus Virchow, ALS Ambulanz, Berlin
  - Neurologische Universitatsklinik Bergmannsheil, Bochum
  - Poliklinik der Universitat Erlangen-Nurnberg, Neurologische Klinik, Erlangen
  - Martin-Luther-Universitat Halle-Wittenberg, Klinikum der Medizinischen Fakultat, Universitatsklinik und Poliklinik fur Neurologie, Halle
  - Medizinische Hochschule Hannover, Neurologische Klinik, Hanover
  - Interdisziplinares Zentrum fur Palliativmedizin, München
  - Klinik und Poliklinik fur Neurologie der Universitat Ulm-Universitatsklinikum Ulm, Ulm
  - Deutsche Klinik fur Diagnostik, Fachbereich Neurologie, Wiesbaden
- Italy (3):
  - Dipartimento di Neurologia e Laboratorio di Neuroscienze - Universita di Milano - IRCCS - Istituto Auxologico Italiano, Milan
  - Divisione di Neuroriabilitazione II - Fondazione Salvatore Maugeri - IRCCS, Pavia
  - Dipartimento di Neuroscienze - Divisione di Neurologia II - Azienda Ospedaliera S. Giovanni Battista - Molinette, Torino
- Netherlands (2):
  - Academic Medical Centre (AMC) Amsterdam - Dept of Neurology, Amsterdam
  - University Medial Center Utrecht, Utrecht
- Kantonsspital St. Gallen, Muskelzentrum/ALS Clinic, Sankt Gallen, Switzerland
- United Kingdom (3):
  - Academic Neuroscience Centre, London
  - Royal Preston Hospital, Preston
  - University of Sheffield - Academic Neurology Unit, Sheffield